CLINICAL TRIAL: NCT05732961
Title: A Phase 2, Single Arm Study of Luspatercept for the Treatment of Anemia in Lower Risk Myelodysplastic Syndromes (MDS) or Non-Proliferative Myelodysplastic Syndromes/ Myeloproliferative Neoplasms (MDS/MPN)
Brief Title: Luspatercept for Anemia in Lower Risk MDS or Non-proliferative MDS/MPN Neoplasms
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-21405
Record Dates: First submitted 2023-02-08; First posted 2023-02-17 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Myelodysplastic Syndromes; Myeloproliferative Neoplasm; Anemia
Keywords: MDS; MPN; Non-Proliferative MDS; Non-Proliferative MPN
MeSH Terms: conditions — Myelodysplastic Syndromes; Myeloproliferative Disorders; Anemia | interventions — luspatercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Participants with gene mutations other than SF3B1 (Experimental): Participants with lower risk MDS or non-proliferative MDS/MPN with somatic splicing gene mutations other than SF3B1
  Interventions: Drug: Luspatercept
- Participants with SF3B1 mutation (Experimental): Participants with lower risk MDS or non-proliferative MDS/MPN with SF3B1 mutation who had received hypomethylating agents and or lenalidomide.
  Interventions: Drug: Luspatercept

INTERVENTIONS:
Drug: Luspatercept — Participants will be treated with Luspatercept, with a starting dose of 1.0 mg/kg subcutaneous injection every 3 weeks (administered on Day 1 of each 21-day treatment cycle)
  Other Names: ACE-536

SUMMARY:
The purpose of the study is to see if participants with anemia due to their type of MDS or MDS/MPN will experience a more decreased need for regular blood transfusions if they take luspatercept plus best supportive care, and what effect, good and/or bad, luspatercept has on them and their anemia due to MDS or MDS/MPN. The safety and tolerability of luspatercept will also be evaluated in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is ≥18 years at the time of signing the informed consent form
2. Participant is willing and able to adhere to the study visit schedule and other protocol requirements
3. Documented diagnosis of MDS or non-proliferative MDS/MPN (WBC < 13,000 U/L)

   1. According to WHO 2016 classification
   2. Meets IPSS-R classification of very low, low, or intermediate risk disease
4. Documented acquired splicing gene mutation

   1. Cohort 1: detectable splicing mutation other than SF3B1: (SRSF2, U2AF1, ZRSR2)
   2. Cohort 2: SF3B1 mutation with prior treatment with hypomethylating agent and or lenalidomide
5. <5% blasts in bone marrow
6. Refractory, intolerant to, or ineligible for, prior ESA treatment, as defined by any one of the following:

   1. Refractory to prior ESA treatment - non-response or response that is no longer maintained. ESA regimen must have been either:

      * rHu EPO ≥ 40,000 IU/wk for at least 8 doses or equivalent Or darbepoetin alpha ≥ 500 μg Q3W for at least 4 doses or equivalent
   2. Intolerant to prior ESA treatment - discontinuation of prior ESA-containing regimen, at any time after introduction due to intolerance or AE
   3. ESA ineligible - Low chance of response to ESA based on endogenous serum EPO > 200 U/L for subjects not previously treated with ESAs
7. Discontinuation of ESAs, G-CSF, GM-CSF ≥ 4 weeks prior to start of study treatment
8. Require RBC transfusions

   a. Average of ≥ 2 units/8 weeks of pRBCs confirmed for a minimum of 16 weeks immediately preceding registration
9. Applies to on treatment subjects only - females of childbearing potential (FCBP) defined as a sexually mature woman who:

   1. has achieved menarche at some point,
   2. has not undergone a hysterectomy or bilateral oophorectomy, or
   3. has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (ie, has had menses at any time in the preceding 24 consecutive months) and must:

      * Have two negative pregnancy tests 48 hours apart as verified by the investigator prior to starting study therapy. She must agree to ongoing pregnancy testing during the course of the study, and after end of study therapy. This applies even if the subject practices true abstinence* from heterosexual contact.
      * Either commit to true abstinence*from heterosexual contact (which must be reviewed on a monthly basis and source documented) or agree to use, and be able to comply with highly effective, contraception without interruption, 35 days prior to starting
10. investigational product (IP), during the study therapy (including dose interruptions), and for 84 days after discontinuation of study therapy
11. Applies to on treatment subjects only - Male subjects must:

    1. Practice true abstinence* (which must be reviewed on a monthly basis) or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions and for at least 84 days following investigational product discontinuation even if he has undergone a successful vasectomy. * True abstinence is acceptable when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception).

Exclusion Criteria:

1. Prior allogeneic or autologous stem cell transplant
2. MDS associated with del 5q cytogenetic abnormality if no prior lenalidomide treatment
3. Uncontrolled hypertension, defined as repeated elevations of diastolic blood pressure (DBP) ≥ 100 mmHg despite adequate treatment
4. ANC < 500/μL (0.5 x 109/L)
5. Platelet count ˂50,000/μL (50 x 109/L)
6. Active other malignancies
7. Severe renal impairment (eGFR < 30 mL/min/1.73 m2)
8. ALT or AST ≥ 3 × ULN
9. Prior treatment with Luspatercept or Sotatercept
10. Pregnant or breastfeeding females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-02-21 (Actual); Primary Completion 2026-06-20 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
RBC Transfusion Independence | From start of treatment to up to 18 months
  RBC transfusion independence (RBC-TI) as defined by IWG 2006 MDS response criteria

SECONDARY OUTCOMES:
Incidence of treatment related adverse events | From start of treatment to 30 days after the last day of treatment, up to 19 months
  To determine the number of participants with treatment related AEs using CTCAE v5
Hematological Improvement | From start of treatment to up to 18 months
  Hematological improvement as defined by using IWG 2006 MDS response criteria
Duration of Response | From start of treatment to up to 18 months
  The duration of response is measured from the time measurement criteria are met for RBC TI or HI by IWG 2006 criteria until the first date of loss of response or progressive disease is objectively documented.
ASC specks changes with response | End of treatment, up to 18 months
  ASC specks as biomarker of response, investigators will compare mean baseline percentage of ASC specks among responders and non-responders (t-test) and use paired t-test to compare change in mean percentage of ASC specks with treatment among responders and non-responders

CONTACTS AND LOCATIONS:
Overall Officials: Rami Komrokji, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided